CLINICAL TRIAL: NCT04163653
Title: Lymphatic Morphology and Classification in Patients With a Fontan Circulation - A Multicenter Study
Brief Title: Lymphatic Morphology of Fontan Patients
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: InCor Heart Institute (Other); Hospital das Clínicas de Ribeirão Preto (Other)
Responsible Party: Sponsor
Other Study IDs: BRALYMF
Record Dates: First submitted 2019-11-11; First posted 2019-11-15 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2021-04

CONDITIONS: Lymphatic Abnormality; Plastic Bronchitis; Protein-Losing Enteropathies; Univentricular Heart; Congenital Heart Disease
MeSH Terms: conditions — Lymphatic Abnormalities; Protein-Losing Enteropathies; Univentricular Heart; Heart Defects, Congenital | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fontan Group: Fontan patients operated at the two centres between 1991 and 2014.
  Interventions: Diagnostic Test: Non-contrast MRI; Diagnostic Test: Cardiopulmonary exercise test
- Healthy Control Group: Age, gender and weight matched healthy controls.
  Interventions: Diagnostic Test: Non-contrast MRI; Diagnostic Test: Cardiopulmonary exercise test

INTERVENTIONS:
Diagnostic Test: Non-contrast MRI — Classification and characterization of the lymphatic vasculature using non-contrast MRI.
Diagnostic Test: Cardiopulmonary exercise test — Cardiopulmonary exercise test, measurement of VO2 and heart rate.

SUMMARY:
The Fontan procedure has revolutionized the treatment of patients born with a congenital univentricular heart defect. However, over time, it is associated with severe lymphatic complications such as plastic bronchitis, protein-losing enteropathy (PLE) and peripheral edema.

The hypothesis is that patients with a univentricular circulation have a changed morphology which may be associated with both the degree of lymphatic complications and their physical capacity.

The morphology will be described using T2-weighted non-contrast MRI.

DETAILED DESCRIPTION:
The Fontan procedure has revolutionized the treatment of patients born with a congenital univentricular heart defect. However, over time, it is associated with severe lymphatic complications such as plastic bronchitis, protein-losing enteropathy (PLE) and peripheral edema. It has been proposed that these complications arise due to a elevated central venous pressure of the changed circulation.

The hypothesis of the study is that patients with a univentricular circulation have a changed morphology which may be associated with both the degree of lymphatic complications and their physical capacity.

The morphology will be described using T2-weighted non-contrast MRI. The main lymphatic vessel, the thoracic duct, will be rendered and measured using 3D software, and the lymphatic changes characterized by Dr. Yoav Dori (CHOP, Pennsylvania, USA), using a newly published grading system. The above will be correlated with the amount of complications experienced by the patients, and their physical capacity measured by both IPAQ questionaire and CPX test.

The study population consists of patients with a Fontan circulation operated at InCor Heart Institute, São Paulo, Brasil and Hospital das Clínicas, Ribeirão Preto, Brasil. Exclusion criteria were mental illness, genetic syndromes and age <18 years. The patient group will be compared with age, gender and weight matched healthy controls.

ELIGIBILITY:
Inclusion Criteria:

- Fontan Circulation

Exclusion Criteria:

* Age <18 years
* Mental illness
* Genetic syndromes

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a Fontan circulation.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Lymphatic classification | 1 hour
  Classified by third party, according to following: (https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6542623/)
Relative measure of tortuosity | 1 hour
  Straight length/full length (mm/mm)
Measurement of thoracic duct volume | 1 hour
  Volume (mm^2)
Measurement of thoracic duct diameter | 1 hour
  Diameter at inlet (mm)
The International Physical Activity Questionnaire (IPAQ-SF) | 1 hour
  IPAQ-SF estimation of weekly activity. (Total Physical Activity min/wk: 2 × time spent on vigorous + moderate + walking) Higher value equals higher level of activity.
CPX heart rate | 1 hour
  Maximum heart rate (bpm)
CPX Vo2 | 1 hour
  VO2 max

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiothoracic and Vascular Surgery, Aarhus N, Denmark